CLINICAL TRIAL: NCT04240366
Title: Additional Left Atrial Appendage Isolation During Balloon Ablation for Persistent or Long-standing Persistent Atrial Fibrillation
Acronym: LALA-LAND-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Principal Investigator, Roland Richard Tilz, MD, Head of Electrophysiology Department, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-323
Record Dates: First submitted 2019-12-18; First posted 2020-01-27 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Persistent or Long-standing Persistent Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Other): Balloon-based ablation of atrial fibrillation by pulmonary vein isolation alone
  Interventions: Procedure: Control intervention
- Group 2 (Experimental): Balloon-based ablation of atrial fibrillation by pulmonary vein and left atrial appendage isolation
  Interventions: Procedure: Experimental intervention

INTERVENTIONS:
Procedure: Control intervention — patients treated with balloon-based ablation of AF by PVI
  Other Names: Balloon-based ablation of atrial fibrillation by pulmonary vein isolation alone
  Arms: Group 1
Procedure: Experimental intervention — patients treated with balloon-based ablation of AF by PVI
  Other Names: Experimental: Group 2 Balloon-based ablation of atrial fibrillation by pulmonary vein and left atrial appendage isolation
  Arms: Group 2

SUMMARY:
Additional left atrial appendage isolation during balloon ablation for persistent or long-standing persistent atrial ﬁbrillation can reduce atrial ﬁbrillation reoccurrence within 3-12 months compared to balloon-based pulmonary vein isolation only.

DETAILED DESCRIPTION:
The intervention in the LALA-LAND-AF trial is the additional LAAI in patients with catheter ablation for persistent AF and will be performed once as index ablation as outlined above. With exception of the index ablation, all patients will be treated according to the current clinical practice guidelines for AF as stated by the European Society of Cardiology (ESC) 11,18 and an expert consensus statement on catheter and surgical ablation1. Patients may be treated with a specific antiarrhythmic drug (AAD) for a maximum of 3 months following the index ablation. No repeat ablation for AF should be performed within the first 3 months. Thereafter, repeat ablations are permitted for recurrent AF irrespective of group allocation. Ablation strategy at repeat ablation includes PV re-isolation if required in both groups and re-isolation of the LAA in the intervention group. In the control group, LAAI may only be performed in case all PV were isolated.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent or long-standing persistent AF (i.e. continuous AF that was/is sustained >7 days or >12 months, respectively)
2. Age ≥18 and ≤80 years
3. Indication for AF ablation as per current guidelines

Exclusion Criteria:

1. Missing informed consent
2. LAA diameter >25mm 10mm distant from circumflex artery assessed by TEE
3. Paroxysmal atrial ﬁbrillation
4. Long-standing persistent atrial ﬁbrillation with a continuous AF duration of >4 years
5. Previous pulmonary vein isolation or MAZE surgery
6. Previous led atrial appendage closure or surgical excision
7. Left atrial diameter >60 mm at baseline
8. Left atrial thrombus at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Time until any documented episode of ATa | 3 - 12 months
  Time until any documented episode of atrial tachyarrhythmia (ATa: atrial fibrillation or atrial tachycardia) lasting longer than 30 seconds within 3-12 months after index ablation without antiarrhythmic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Roland R. Tilz, Prof. Dr., Study Director — Universitätsklinikum Schleswig-Holstein, Universitäres Herzzentrum Lübeck, Klinik für Rhythmologie; Sorin S. Popescu, MD, Study Chair — Universitätsklinikum Schleswig-Holstein, Universitäres Herzzentrum Lübeck, Klinik für Rhythmologie
Locations (3):
- Germany (3):
  - University Hospital Eppendorf, Hamburg, Germany, Hamburg, Hamburg
  - Asklepios Klinik Altona, Hamburg, Hamburg
  - Clinic for Rhythmologiy Luebeck, Schleswig-Holstein Germany, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No